CLINICAL TRIAL: NCT02923765
Title: Efficacy of Stepper Aerobic Training on Cardiopulmonary Fitness, Disability, Systemic Inflammation and Thrombosis in Stroke Patients With Hemiplegia
Brief Title: Stepper Aerobic Training on Fitness, Disability, Inflammation and Thrombosis in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201601026B0
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2020-02

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- combined training (CT) (Active Comparator): additional aerobic training by a stepper : 35 minutes/session, 5 sessions/week and 4-5 weeks
  Interventions: Other: Aerobic training by a stepper
- usual rehabilitation (UR) (No Intervention): Usual rehabilitation, without additional aerobic training
- healthy participant (HP) (No Intervention): healthy control

INTERVENTIONS:
Other: Aerobic training by a stepper — Aerobic training by a stepper: 35 minutes/session, 5 sessions/week and 4-5 weeks in total
  Arms: combined training (CT)

SUMMARY:
Stroke rehabilitation of hemiplegics primarily lies in motor control and training of activities of daily life. Whole body aerobics is much less emphasized. Nonetheless, cardiopulmonary fitness of even ambulatory hemiparetics is only half compared with healthy people, which is prone to deconditioning. The present study aims to understand the efficacy of aerobic training in addition to the usual neuro-rehabilitation, including aerobic fitness, daily activities dependency, anti-inflammation and anti-thrombosis. This is a prospective and randomized design. The subjects will be recruited from the hospitalized patients in the rehabilitation ward of Chang Gung Memorial Hospital at Linkuo. 120 hemiplegic patients due to stroke will be enrolled and randomized into two groups: combined training (CT) and usual rehabilitation. Participants in CT will receive aerobics at moderate intensity in addition to the usual rehabilitation. The program has 35 minutes/session, 5 sessions/week and 4-5 weeks in total. A constant-power semi-recumbent stepper will be employed as the training modality. It uses bilateral reciprocal movement of the arm coupled with the opposite leg, which allows for a push and pull motion. Additional 20 healthy participants will also be recruited as the healthy control. Assessment before and after training includes: (I) graded cardiopulmonary exercise test using constant-load stepper. (II) Functional Independence Measure. (III) coagulation system assessment, using Thrombin generation assay and Ceveron alpha (Technoclone GmbH, Vienna, Austria) : Von Willebrand factor, tissue plasminogen activator, plasminogen activator inhibitor-1, D-dimer, factor VIII, etc. [the 1st year]; (IV) monocyte-platelet aggregation and its subtypes, using flow cytometry [the 2nd year]. ( V) systemic inflammation, platelet activation and prognostic biomarker：C-reactive protein, soluble P-selectin, asymmetric dimethylarginine, Lipoprotein-Associated Phospholipase A2, etc [the 3rd year]. Statistical analysis will use ANOVA with post-hoc, two-way repeated measure ANOVA, etc. The investigation will start after approval and end in 2019, July. We hope this investigation will establish a more comprehensive rehabilitation program for clinical application.

DETAILED DESCRIPTION:
In Taiwan, there are 220,00 stroke survivors and each year, 10,000 new suffers causing impairment in daily activities. This is the leading cause of disability and consumes 4.5 billions of National Health Insurance yearly. More than half of them become hemi-paretics and hemi-plegics. Stroke leads to the adverse combination of reduced functional capacity and increased energy demands to perform routine activities Thereby, physiologic fitness reserve is diminished. Aerobic fitness is low in stroke survivors. Among ambulatory patients suffering from hemiparetic stroke, the VO2peak is approximately half that of age-matched individuals , a level that is near the minimum range required for activities of daily life. It may limit their ability to perform everyday activities and cause further complications, such as cardiopulmonary de-conditioning, muscular atrophy, joint stiffness, or even learned nonuse.

Many patients are discharged from neurorehabilitation focusing on motor control and ADL (activity of daily life ) training, while aerobic fitness training is neglected, especially in non-ambulatory patients. Randomized exercise training studies using a wide variety of modalities and protocols have demonstrated an 8~23% improvement in VO2peak after 2-6 months of training . However, most research recruit patients with hemiparesis who have mild-to-moderate gait impairment . No specific training protocols has been adequately studied or can be suggested for hemiplegic patients. It is difficult for them to partake in aerobic exercise, like walking or biking. There is a need to develop a new aerobic exercise module suitable for the patients, especially for those with ambulation difficulty resulted from severe paralysis.

In the current investigation, a semi-recumbent stepper with constant power design will be adopted as training modality. It accommodates motor function deficits by providing trunk and distal limb support . In addition, semi- recumbent stepper uses bilateral reciprocal movement of the arm coupled with the opposite leg, which allows for a push and pull motion.

Aerobic fitness training has been proposed as a beneficial approach for people with stroke. Taking part in fitness training could have a range of other benefits important to people with stroke such as improving cognitive function, improving mood, and quality of life, and it could reduce the risk of recurrent stroke . In the present investigation, the outcome measurement will not only include cardiopulmonary fitness and the degree of daily activity dependency, but also prognostic biomarkers, thrombotic and inflammatory state.

It is well-documented that exercise training has an anti-thrombotic effect . Increased physical activity and cardiorespiratory fitness are associated with a reduced risk of fatality from cardiovascular diseases. Moreover, increased studies have demonstrated that regular moderate-intensity physical activity is associated with health benefits, even when aerobic fitness (e.g., maximal oxygen uptake, VO2max) remains unchanged . For sedentary persons at risk for cardiovascular disease, adopting a moderately active lifestyle can induce important health benefits, such as reducing prothrombotic factors and lipid peroxidation , increasing fibrinolytic activity and high-density lipoprotein levels , etc. One of the present investigation aims to understand whether 20~25 sessions of aerobic training at moderate intensity will induce these favorable adaptations that could contribute to decreased risk for ischemic event.

This is a prospective randomized controlled study. Eighty stroke sufferers with unilateral weakness will be enrolled in Chang Gung Memorial Hospital at Linkuo. They will be randomized into two groups: combined training (CT) and usual rehabilitation (UR). Participants in the CT group will receive supervised aerobic training at moderate intensity in addition to usual neuro-rehabilitation, in which motor control and task-oriented ADL training are the major contents. Patients in the UR will undergo usual neuro-rehabilitation only. The aim of the present research is to evaluate the efficacy of an aerobic training program at moderate intensity for a total of 20~25 sessions using a semi-recumbent stepper with constant power design. Pre- and post-training measurement includes (I) cardiopulmonary fitness, (II) daily activities dependency, (III) coagulation and fibrinolysis profile. [the 1st year] (IV) monocyte subsets and its interaction with platelets [the 2nd year]. (V) Systemic inflammation, platelet activation and prognostic biomarker：C-reactive protein, soluble P-selectin, asymmetric dimethylarginine, Lipoprotein-Associated Phospholipase A2, etc. [the 3rd year]. Venous blood will be sampled two times before and after rehabilitation.

Hopefully, this clinical investigation will establish the model of incorporating aerobics in the hemiplegic patients following stroke, and its efficacy for clinical application.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ischemic stroke
* Must be able to ride the stepper
* No cardiovascular disease in the healthy control group

Exclusion Criteria:

* Resting heart rate greater than 100 beats per minute
* Atrial fibrillation or flutter
* Poor control of high blood pressure or diabetes
* Patients with peripheral arterial occlusive disease
* Patients with end-stage renal disease
* Patients receiving anticoagulant therapy
* Neurological instability
* Confusion or cognitive dysfunction

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Exercise capacity of all participants by Cardiopulmonary ExerciseTest (CPET) and Functional Independence Measure (FIM) | three years
  CPET

SECONDARY OUTCOMES:
Thrombosis and Coagulation Activities of Blood Samples of All Participants by Flow Cytometry, | three years
  detection of monocytes and platelets aggregation
Thrombosis and Coagulation Activities of Blood Samples of All Participants by Dynamic TG Assay | three years
  detection the amount and time of thrombin generation.
Thrombosis and Coagulation Activities of Blood Samples of All Participants Enzyme-linked Immunosorbent Assay (ELISA) | three years
  ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Chun Huang, MD, PhD, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Shu-Chun Huang, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No